CLINICAL TRIAL: NCT03643068
Title: Phase 1A Study of the Safety of KSP/QRH Dimer in Humans for the Early Detection of GI Malignancies
Brief Title: Phase 1A Study of the Safety of KSP/QRH Dimer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Danielle Kim Turgeon, Professor of Internal Medicine, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00141420
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Peptides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KSP-QRH-E3-IRDye800 (Peptide 919288G) 0.6 mg subjects 1-3 (Experimental): The first three subjects will receive lyophilized powder reconstituted with 5 mL of 0.9% NaCl, 0.6 mg of KSP-QRH-E3-IRDye800 (Peptide 919288G) total. For the first three subjects, 3.34 mL of KSP-QRH-E3-IRDye800 (Peptide 919288G)will be discarded. The 1.66 mL of KSP-QRH-E3-IRDye800 (Peptide 919288G)remaining in the syringe will be administered by squirting it into the mouth of the subject.
  Interventions: Drug: KSP-QRH-E3-IRDye800 (Peptide 919288G), 0.6 mg
- KSP-QRH-E3-IRDye800 (Peptide 919288G) 1.8 mg subjects 4-25 (Experimental): Following a safety review of the first three subjects receiving 0.6 mg dose, the remaining 22 subjects will receive the full 1.8 mg dose of KSP-QRH-E3-IRDye800 (Peptide 919288G) reconstituted in 5 mL 0.9% NaCl. These 22 subjects will receive all 5 mL of the peptide solution in a syringe for administration. The agent will not be reconstituted until the subject is ready to squirt the peptide into his or her mouth via syringe. They will be asked to wait 5 minutes and then drink at least 4-8 oz of tap water.
  Interventions: Drug: KSP-QRH-E3-IRDye800 (Peptide 919288G), 1.8 mg

INTERVENTIONS:
Drug: KSP-QRH-E3-IRDye800 (Peptide 919288G), 0.6 mg — The investigational agent to be used in this study is KSP/QRH dimer: a fluorescently-labeled peptide dimer composed of a 14-amino acid sequence [Lys-Ser-Pro-Asn-Pro-Arg-Phe] and [Gln-Arg-His-Lys-Pro-Arg-Glu] attached via a PEG3, Lys and Cys linker [PEG3]2-Lys-Cys to a near-infrared fluorophore, IRDye800CW (0.6 mg dose).
  Arms: KSP-QRH-E3-IRDye800 (Peptide 919288G) 0.6 mg subjects 1-3
Drug: KSP-QRH-E3-IRDye800 (Peptide 919288G), 1.8 mg — The investigational agent to be used in this study is KSP/QRH dimer: a fluorescently-labeled peptide dimer composed of a 14-amino acid sequence [Lys-Ser-Pro-Asn-Pro-Arg-Phe] and [Gln-Arg-His-Lys-Pro-Arg-Glu] attached via a PEG3, Lys and Cys linker [PEG3]2-Lys-Cys to a near-infrared fluorophore, IRDye800CW (1.8 mg dose).
  Arms: KSP-QRH-E3-IRDye800 (Peptide 919288G) 1.8 mg subjects 4-25

SUMMARY:
To evaluate the safety of orally administered KSP-QRH-E3-IRDye800 (Peptide 919288G), a topically administered Li-Cor IRDye800CW labeled heptapeptide dimer (KSP/QRH Dimer) specific for human epithelial growth factor receptor 2 (HER2) and epidermal growth factor receptor (EGFR).

DETAILED DESCRIPTION:
This is a Phase IA study of the safety of an orally administered KSP-QRH-E3-IRDye800 (Peptide 919288G) heptapeptide dimer for detection of neoplastic tissues in multiple areas of the gastrointestinal tract in humans. The investigators intend to enroll 25 evaluable subjects. The investigators expect to be able to enroll about 2-3 subjects per week, so the study should take about 2-3 months to complete.

Interested, healthy subjects ages 25-100 who respond to recruitment advertising on UMHealthResearch.org and appear to be eligible based responses to inclusion/exclusion criteria questions will be scheduled for a study visit at MCRU. At the study visit, the subjects will review and sign the informed consent and eligibility will be confirmed. If eligible, subjects will provide a blood sample for clinical labs and a urine sample for urinalysis, as well as have an EKG. A negative urine pregnancy test for women of child-bearing potential is required to be eligible. Eligible subjects will consume the reconstituted KSP-QRH-E3-IRDye800 (Peptide 919288G). After 5 minutes, subjects will drink a minimum 4-8 ounces of tap water and vital signs will be taken. Subjects will remain in MCRU for observation for 30 minutes. Vital signs will be recorded after 30 minutes, and another EKG will be conducted. Subjects are required to return to MCRU to have a repeat blood draw for clinical labs and urinalysis within 24 to 48 hours after KSP-QRH-E3-IRDye800 (Peptide 919288G) ingestion. The study team will conduct a verbal assessment for toxicity at this visit.

ELIGIBILITY:
Inclusion Criteria:

* Not pregnant (willing to have pregnancy test if applicable)
* No recent illness (infection, URI, virus or flu) within 2 weeks,
* Stable health status (i.e. no medication changes within 2 months, no recent surgery, etc. per PI)
* Willing and able to sign informed consent
* Willing and able to drink the peptide and a tap water chaser
* Willing and able to get baseline and 24-48 hours post ingestion labs
* Willing and able to get pre and post ingestion EKG

Exclusion Criteria:

* Known allergy to li-cor IRDye800CW, a near infrared fluorosphore or derivatives
* Subjects on active chemotherapy or radiation therapy
* Diabetics on insulin/hypoglycemic (due to fasting requirements)

Ages: 25 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2018-10-27 (Actual); Study Completion 2018-10-27 (Actual)

PRIMARY OUTCOMES:
Number of subjects with abnormal lab values | 48 hours
  review of laboratory values for abnormalities after intervention with KSP/QRH Dimer
Number of subjects with unexpected side effects | 48 hours
  Side effects collected through their follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Chandhrasekhar, BS, Study Chair — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States